CLINICAL TRIAL: NCT07367503
Title: Investigation of the Role of Systemic Immune-Inflammatory Index in Spontaneously Regressing Lumbar Disc Hernias
Brief Title: SIII and Spontaneous Regression in Lumbar Disc Herniation
Acronym: SIII-LDH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Çanakkale Onsekiz Mart University (Other)
Responsible Party: Principal Investigator, Ali Akar, Assoc. Prof., Çanakkale Onsekiz Mart University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: COMU-BS-1; THD-2023-4339 (Other Grant/Funding Number: Çanakkale Onsekiz Mart University's Scientific Research Coordination Unit)
Record Dates: First submitted 2026-01-18; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Inflammation; Neutrophil; Lymphocyte; Neurosurgery
Keywords: Inflammation; neutrophil; lymphocyte; neurosurgery
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (No Intervention): No intervention the group and healty
- Surgical treatment group (Other): Already operated
  Interventions: Other: Lumbar disc herniation surgery
- Medical treatment group (Other): Already have a treatment protocol
  Interventions: Other: Lumbar disc herniation treatment

INTERVENTIONS:
Other: Lumbar disc herniation treatment — Lumbar disc herniation medical treatment
  Arms: Medical treatment group
Other: Lumbar disc herniation surgery — Lumbar disc herniation surgecal treatment
  Arms: Surgical treatment group

SUMMARY:
This study aimed to investigate the role of the Systemic Immune-Inflammatory Index (SIII) in patients with lumbar disc herniation (LDH) and to evaluate its potential clinical relevance in relation to treatment modality.

DETAILED DESCRIPTION:
Lumbar disc herniation (LDH) is a common spinal disorder that may be managed conservatively or surgically depending on clinical severity and response to treatment. Inflammatory and immune-mediated mechanisms are known to contribute to disc degeneration and symptom progression; however, reliable and easily accessible biomarkers that may assist in treatment decision-making remain limited. The Systemic Immune-Inflammatory Index (SIII), derived from peripheral blood neutrophil, platelet, and lymphocyte counts, has emerged as a comprehensive indicator reflecting systemic inflammatory and immune status.

This retrospective observational study evaluated patients diagnosed with lumbar disc herniation who were followed in the Neurosurgery Clinic between June 1, 2020, and January 30, 2023. Demographic characteristics, clinical and neurological findings at admission, comorbidities, treatment modality, laboratory parameters, and radiological findings were obtained from medical records. Patients were categorized into three groups: those managed conservatively with medical treatment, those who underwent surgical intervention, and healthy individuals included as a control group.

Peripheral blood parameters, including neutrophil and lymphocyte counts, were recorded, and the neutrophil-to-lymphocyte ratio (NLR) and SIII values were calculated. Comparisons of inflammatory markers were performed among the medical treatment, surgical treatment, and control groups to assess differences related to disease severity and treatment approach.

The analysis demonstrated significantly higher neutrophil counts, NLR, and SIII values in patients who required surgical treatment compared with both medically treated patients and healthy controls. These findings indicate that elevated systemic inflammatory indices are associated with more severe clinical presentations requiring surgical intervention.

Overall, this study aims to clarify the clinical relevance of SIII in lumbar disc herniation and to explore its potential role as an adjunct biomarker for evaluating disease severity and supporting treatment decisions in routine clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Dagnosis of lumbar disc herniation confirmed by magnetic resonance imaging (MRI)
* Follow-up at the Department of Neurosurgery between June 1, 2020, and January 30, 2023
* Availability of baseline complete blood count and inflammatory marker data
* For the surgical group: Patients who underwent single-level, unilateral lumbar microdiscectomy (LMD) for acute lumbar disc herniation
* For the medical treatment group: Patients with single-level, unilateral lumbar disc herniation who did not undergo surgery and demonstrated spontaneous regression during follow-up after medical treatment
* For the control group: Individuals without spinal disease who applied to the outpatient clinic with headache complaints and had available routine blood test results

Exclusion Criteria:

* Previous medical or surgical treatment for lumbar disc pathology
* Presence of systemic inflammatory disease
* Rheumatic disease
* Tumoral or malignant pathology
* History of spinal trauma
* Active infection at the time of blood sampling
* Congenital spinal anomalies
* Incomplete clinical, laboratory, or radiological data

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2023-01-30 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
Systemic Immune-Inflammatory Index (SIII) | At baseline (at initial diagnosis)
  Calculated from peripheral blood neutrophil, platelet, and lymphocyte counts.

CONTACTS AND LOCATIONS:
Locations (1):
- Çanakkale Onsekiz Mart University, Çanakkale, Center, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Oliveira CB, Maher CG, Pinto RZ, Traeger AC, Lin CWC, Chenot JF, et al. Clinical practice guidelines for the management of non-specific low back pain in primary care: an updated overview. European Spine Journal [Internet]. 2018 Nov 1 [cited 2024 Apr 29];27(11):2791-803. Available from: https://link.springer.com/article/10.1007/s00586-018-5673-2 2. Hoy D, March L, Brooks P, Blyth F, Woolf A, Bain C, et al. The global burden of low back pain: estimates from the Global Burden of Disease 2010 study. Ann Rheum Dis [Internet]. 2014 Jun 1 [cited 2024 Apr 29];73(6):968-74. Available from: https://ard.bmj.com/content/73/6/968 3. Lagerbäck T, Fritzell P, Hägg O, Nordvall D, Lønne G, Solberg TK, et al. Effectiveness of surgery for sciatica with disc herniation is not substantially affected by differences in surgical incidences among three countries: results from the Danish, Swedish and Norwegian spine registries. Eur Spine J [Internet]. 2019 Nov 1 [cited 2024 Apr 29];28(11):2562-71. Available from: https://pubmed.ncbi.nlm.nih.gov/30269234/ 4. Johansen JG. Demonstration of anterior intervertebral disc herniation by CT. Neuroradiology. 1987 Mar;29(2):214. 5. Teplick JG, Haskin ME. Spontaneous regression of herniated nucleus pulposus. AJR Am J Roentgenol [Internet]. 1985 [cited 2024 Apr 29];145(2):371-5. Available from: https://pubmed.ncbi.nlm.nih.gov/3875236/